CLINICAL TRIAL: NCT02424539
Title: A Randomized, Doubled-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Once-Daily, Intranasal Administration of Fluticasone Furoate Nasal Spray 55 mcg and 110 mcg for 4 Weeks in Chinese Pediatric Subjects Ages 2 to 12 Years With Allergic Rhinitis
Brief Title: A Study to Compare the Efficacy and Safety of Fluticasone Furoate Nasal Sprays (FFNS) 55 Microgram (mcg) and 110 mcg in Chinese Pediatric Subjects With Allergic Rhinitis (AR)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201492
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-12

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal; Rhinitis, Allergic
Keywords: Seasonal; Fluticasone Furoate; Perennial; Allergic Rhinitis; Nasal Spray
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FFNS 55 mcg Arm (Experimental): Each subject will be dispensed with two nasal spray device labelled as Device A and Device B containing either FF or Placebo. Subject's on their own or with assistance from parent/guardian will administer FFNS 55 mcg per day, one intranasal spray from Device A, once daily into each nostril (27.5 mcg per spray) and another spray of placebo nasal spray from Device B, once daily into each nostril, in the morning for 4 Weeks.
  Interventions: Drug: FFNS; Other: Placebo
- FFNS 110 mcg Arm (Experimental): Each subject will be dispensed with two nasal spray device labelled as Device A and Device B containing FF or Placebo. Subject's on their own or with assistance from parent/guardian will administer FFNS 110 mcg per day, one intranasal spray from Device A, once daily into each nostril (27.5 mcg per spray) and another spray of placebo nasal spray from Device B, once daily into each nostril, in the morning for 4 Weeks.
  Interventions: Drug: FFNS; Other: Placebo
- Placebo Arm (Placebo Comparator): Each subject will be dispensed with two nasal spray device labelled as Device A and Device B containing only placebo. Subject's on their own or with assistance from parent/guardian will administer one intranasal spray of placebo, from Device A and Device B, once daily into each nostril in the morning for 4 Weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FFNS — FF as a aqueous suspension for intranasal inhalation with unit dose strength of 27.5 mcg per dose administered via a metered side-actuated nasal spray device.
  Arms: FFNS 110 mcg Arm; FFNS 55 mcg Arm
Other: Placebo — Placebo as a aqueous suspension to match the other study treatments minus the active component(s) for intranasal inhalation administered via a metered side-actuated nasal spray device.

SUMMARY:
This Phase IV interventional study is a multi-center, randomized, double-blind, placebo-controlled parallel study to evaluate the efficacy and safety of FFNS110 mcg and 55 mcg once daily versus vehicle placebo aqueous nasal spray in chinese pediatric subjects ages 2 to 12 years with AR.

This study comprises screening and run-in period (4 to14 days), double-blind treatment period (28 days) and follows up period (3 to7 days). Subjects entering the study will participate for maximum of 50 days, including five clinical visits and a follow-up contact.

The study is planned to enroll approximately 360 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained from the subject's parent/guardian.
* Chinese male or non-child bearing potential female pediatric outpatients subjects who are >=2 to <=12 years of age at Visit 2.
* Diagnosis of AR: Subjects must have a diagnosis of intermittent allergy rhinitis (IAR) [symptoms are present <4 days a week, or for <4 weeks] or persistent allergic rhinitis (PER) [symptoms are present >=4 days a week, or for >=4 weeks] by symptoms, physical signs skin prick test (SPT) and serum-specific immunoglobulin E (IgE) test. Subjects must have 2 or more symptoms of AR (watery rhinorrhea, nasal obstruction, nasal itching and sneezing), which are also present consecutively or accumulatively more than 1 hour on each day prior to Visit 1, or/and concomitant ocular symptoms: ocular itching, red eyes, watery eyes etc. The physical signs includes: nasal mucosa pale, oedema, nasal secretion. Allergic shiner and allergic crease in severity pediatric. A documented positive prick skin test and a positive serum specific IgE test using standardized allergen extract. A positive skin test is defined as a allergen wheal >=3 millimeters (mm), a histamine >=3 mm. Subjects have nasal symptoms described above or/and associated with ocular symptoms, as well as the nasal signs and one of laboratory test positive or demonstrate SPT represented a positive response or serum-specific IgE testing represented a positive response within 12 months prior to Visit 1.
* Subject must be willing to maintain same environment throughout the study.
* Subject and/or subject's parent/guardian understands and is willing, able and likely to comply with study procedures and restrictions as well as manage study drug administration.

Exclusion Criteria:

* Concomitant Medical Conditions: (a) Significant concomitant medical conditions defined as historical or current evidence of clinically significant uncontrolled disease of any body system. Significant is defined as any disease that, in the opinion of the investigator, would confound the interpretation of the study results if the disease/condition exacerbated during the study: significant renal impairment, which based on the opinion of the investigator, would preclude the subjects' participation in the study and current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). (NOTES: Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis and Chronic stable hepatitis B and C [e.g., presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment] are acceptable if subject otherwise meets entry criteria). (b) A severe physical obstruction of the nose (e.g., deviated septum or nasal polyp) or frequent bleeding of the nose that could affect the deposition of double blind intranasal study drug. (c) Current or history of a Candida infection of the nose or oropharynx, shingles, chickenpox, measles, ocular herpes simplex. (d) Known hypersensitivity to corticosteroids or any excipients in the product. (e) Recent nasal septal surgery or nasal septal perforation. (f) Subjects start, discontinue or change desensitization treatment within 30 days prior to Visit 1. (g) Bacterial or viral infection of the eyes or upper respiratory tract within two weeks of Visit 1 or during the screening period. (h) Asthma, with the exception of mild intermittent asthma. (i) Diagnosis of rhinitis medicamentosa, vasomotor AR or eosinophil rhinitis.
* Abnormal Laboratory Findings: A clinically significant laboratory abnormality including Liver Function Tests at Visit 1 meeting the following criteria: Alanine aminotransferase (ALT) >2 x upper limit of normal (ULN) and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Abnormal Electocardiogram (ECG): Clinically significant abnormal ECG finding at Visit 1. Significant is defined as: Corrected QT (QTc) > 450 milliseconds (msec) or QTc > 480 msec in subjects with Bundle Branch Block. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trail.
* Concomitant Medication: Use of prescription or over-the-counter medication that would significantly affect the course of AR, or interact with study drug, such as: Chronic use of concomitant medications such as tricyclic antidepressants, that would affect assessment of the effectiveness of the study drug; Chronic use of long- acting beta2-agonists (e.g., salmeterol); Potent Cytochrome P450 subfamily enzyme 3A4 [CYP3A4] inhibitors (e.g., ritonavir, ketoconazole, itraconazole, clarithromycin, etc); Allergen immunotherapy for the treatment of allergies.
* Use of followings medications are not allowed throughout the study: Short-acting antihistamines, including ocular preparations and antihistamines contained in anti-cold medicine, insomnia or antalgic; Oral or inhaled anticholinergics; Oral or intranasal decongestants; Oral or intranasal antileukotrienes; Oral or inhaled long-acting beta2 agonists; Chinese traditional medicines that have potential effect to AR; Liquorice preparation; Medications that significantly inhibit the CYP3A4, including ritonavir and ketoconazole; tricyclic antidepressants; long-acting antihistamines( eg. desloratadine, fexofenadine, cetirizine and loratadine [ taken as rescue medication]); Intranasal antihistamines; or Intranasal or ocular cromolyh; Intranasal corticosteroids includes: Inhaled, oral, intramuscular, intravenous, ocular and/or dermatological corticosteroid (with the exception of hydrocortisone cream/ointment, 1% or less) and Immunosuppressive medications; Subcutaneous omalizumab.
* Subjects will travel more than 48 hours during the study may cause the change of allergen.
* Subjects, who, in the opinion of the Investigator or sub-investigators, are not able to comply with the protocol requirements.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 358 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- China (12):
  - GSK Investigational Site, Xiamen, Fujian
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Wenzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20743

REFERENCES:
- [Background] Zhang Y, Wei P, Chen B, Li X, Luo X, Chen X, Xiang M, Li L, Zhao S, Xiao X, Yang X, Chen J, Fu Y, Xiao S, Liu H, Cheng L, Yao H. Intranasal fluticasone furoate in pediatric allergic rhinitis: randomized controlled study. Pediatr Res. 2021 May;89(7):1832-1839. doi: 10.1038/s41390-020-01180-0. Epub 2020 Oct 2. PMID 33007780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This efficacy and safety study of fluticasone furoate (FF) was conducted at 16 centers in China. A total of 505 pediatric participants with allergic rhinitis were screened; of which 147 were screen and run-in failures and 358 were randomized in a 1:1:1 ratio to receive placebo, FF 55 micrograms (µg) or FF 110 µg once daily (QD).
Groups:
- Placebo: Participants received one spray of placebo from nasal spray device A (placebo nasal spray) followed by one spray from nasal spray device B (placebo nasal spray) into each nostril QD in the morning for 28-day treatment period.
- FF 55 µg QD: Participants received one spray of FF 55 µg from nasal spray device A (FF nasal spray) followed by one spray from nasal spray device B (placebo nasal spray) into each nostril QD in the morning for 28-day treatment period.
- FF 110 µg QD: Participants received one spray of FF 110 µg from nasal spray device A (FF nasal spray) followed by one spray from nasal spray device B (FF nasal spray) into each nostril QD in the morning for 28-day treatment period.
Period: Overall Study
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Started | 120 | 119 | 119
Completed | 106 | 111 | 111
Not Completed | 14 | 8 | 8
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 0
Not completed — Other: Reached stopping criteria | 11 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD | Total
Number analyzed (Participants) | 120 | 119 | 119 | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.8 (2.64) | 6.9 (2.54) | 6.6 (2.54) | 6.8 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 32 | 112
  Male | 78 | 81 | 87 | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 120 | 119 | 119 | 358

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daily, Reflective Total Nasal Symptom Scores (rTNSS) Over the First 2 Weeks Treatment Period
Description: TNSS is a composite score of the four components (nasal congestion, itching, rhinorrhea and sneezing) with a total score of 0 to 12. A higher score means a worse nasal symptom. The score of each component ranges from 0 (no symptom) to 3 (severe symptoms). Participants were instructed to provide scores in a reflective manner using their diary. The daily rTNSS was the average of the morning rTNSS and evening rTNSS assessments. The daily scores were averaged to calculate the overall/total score. The morning reflective assessment was performed prior to administering the morning dose. The evening reflective assessment was performed approximately 12 hours after dosing but before bedtime. Baseline scores obtained over "4 days prior to randomization" were average of the last 8 rTNSS assessments (4 AM assessments, 4 PM assessments) over the consecutive four 24-hours periods prior to randomization. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and up to Week 2
Population: Intent-To-Treat (ITT) Population comprised of all randomized participants who received at least one dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Scores on a scale | -1.95 (0.16) | -3.18 (0.16) | -3.28 (0.16)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.68 to -0.78] — Least square (LS) mean difference between placebo and FF 55 µg QD has been presented using analysis of co-variance (ANCOVA) model adjusted for treatment, Baseline value, gender, age and type of Allergic Rhinitis
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.32, 95% CI 2-sided [-1.77 to -0.87] — LS mean difference between placebo and FF 110 µg QD has been presented using ANCOVA model adjusted for treatment, Baseline value, gender, age and type of Allergic Rhinitis

2. Secondary Outcome: Number of Participants Showing Response to the Therapy After the First 2 Weeks Treatment on a 7-point Categorical Scale
Description: Response was defined as effectiveness of study medication for relieving allergic rhinitis symptoms over the entire treatment period. Overall response to therapy was evaluated using the 7-point categorical scale ranging from 1 (significantly improved) to 7 (significantly worse). Number of participants showing response to therapy after the first 2 weeks have been presented. Only those participants with response to therapy over the entire treatment period were included in the analysis.
Time Frame: Week 2
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 113 | 114 | 119
Participants
  Significantly improved | 13 | 38 | 51
  Moderately improved | 30 | 48 | 33
  Mildly improved | 45 | 22 | 29
  No change | 21 | 4 | 4
  Mildly worse | 3 | 1 | 1
  Moderately worse | 1 | 1 | 0
  Significantly worse | 0 | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.24, 95% CI 2-sided [0.14 to 0.39] — Odds ratio for FF 55 µg QD versus placebo has been presented using a logistic regression model with Wald's test with treatment, gender, age and type of Allergic Rhinitis as factors
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.12 to 0.33] — Odds ratio for FF 110 µg QD versus placebo has been presented using a logistic regression model with Wald's test with treatment, gender, age and type of Allergic Rhinitis as factors

3. Secondary Outcome: Mean Change From Baseline of Intranasal Finding Score by Anterior Rhinoscopy at the First 2 Weeks
Description: The nasal concha mucosa symptoms score was used to evaluate change in anterior rhinoscopy. It is a composite score of four components including swelling of inferior nasal concha mucosa, color of inferior nasal concha mucosa, watery secretion volume and description of rhinorrhea. Severity of each of the component was assessed using the scale ranging from 0 (no symptom) to 3 (severe). The 4 components were averaged to obtain a total score which ranges from 0 to 12 where a higher score means a worse nasal symptom. Baseline was defined as 4 days prior to randomization, including the morning symptom assessment on the randomization date. Change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available at the specified time points were included in the analysis.
Time Frame: Baseline and up to Week 2
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 114 | 113 | 117
Scores on a scale | -2.32 (0.25) | -4.47 (0.25) | -4.30 (0.24)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.15, 95% CI 2-sided [-2.84 to -1.46] — LS mean difference between placebo and FF 55 µg QD has been presented using ANCOVA model adjusted for treatment, Baseline value, gender, age and type of Allergic Rhinitis
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.98, 95% CI 2-sided [-2.66 to -1.29] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Mean Change From Baseline Over the First 2 Weeks in the Daily, Reflective Total Ocular Symptoms Score (rTOSS)
Description: TOSS is a composite score of the three components (eye itching and burning, eye watering and eye redness) with a total score of 0 to 9. Higher score means a worse symptom. The score of each component ranges from 0 (no symptom) to 3 (severe symptoms). The daily scores were averaged to calculate the overall/total score. Participants were instructed to provide scores and document their symptoms in a reflective manner twice daily using their diary at the same time of reflective nasal symptoms assessment. Baseline scores obtained over "4 days prior to randomization" were average of the last 8 rTNSS assessments (4 AM assessments, 4 PM assessments) over the consecutive four 24-hours periods prior to randomization. Change from Baseline was defined as post-dose visit value minus Baseline value
Time Frame: Baseline and up to Week 2
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Scores on a scale | -1.15 (0.10) | -1.24 (0.10) | -1.40 (0.10)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p = 0.503, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.38 to 0.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p = 0.078, ANCOVA; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.53 to 0.03] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Mean Change From Baseline in Rescue Loratadine Use (Mean Rescue-free Days) Over the First 2 Weeks Treatment Period
Description: Loratadine was provided as a rescue medication to use if needed throughout the study treatment period. Participants were asked to document loratadine rescue medication use on the daily treatment diary. Baseline was defined as 4 days prior to randomization, including the morning symptom assessment on the randomization date. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and up to Week 2
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Days | 12.76 (0.18) | 13.28 (0.18) | 13.43 (0.18)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p = 0.048, ANCOVA; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [0.01 to 1.02] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = 0.66, 95% CI 2-sided [0.16 to 1.17] — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Mean Change From Baseline in Daily rTNSS Over the 4 Weeks Treatment Period
Description: as for outcome 1
Time Frame: Baseline and up to Week 4
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Scores on a scale | -2.57 (0.17) | -3.93 (0.17) | -4.03 (0.17)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.36, 95% CI 2-sided [-1.83 to -0.90] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.46, 95% CI 2-sided [-1.92 to -0.99] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Number of Participants Showing Response to the Therapy After 4 Weeks Treatment on a 7-point Categorical Scale
Description: Response was defined as effectiveness of study medication for relieving allergic rhinitis symptoms over the entire treatment period. Overall response to therapy was evaluated using the 7-point categorical scale ranging from 1 (significantly improved) to 7 (significantly worse). Number of participants showing response to therapy after the first 4 weeks have been presented. Only those participants with response to therapy over the entire treatment period were included in the analysis.
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 106 | 111 | 111
Participants
  Significantly improved | 22 | 59 | 63
  Moderately improved | 31 | 34 | 34
  Mildly improved | 31 | 13 | 11
  No change | 19 | 4 | 3
  Mildly worse | 1 | 0 | 0
  Moderately worse | 1 | 0 | 0
  Significantly worse | 1 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.20, 95% CI 2-sided [0.12 to 0.34] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.10 to 0.29] — [estimate comment as in outcome 2, analysis 2]

8. Secondary Outcome: Mean Change From Baseline of Intranasal Finding Score by Anterior Rhinoscopy at the First 4 Weeks
Description: as for outcome 3
Time Frame: Baseline and up to Week 4
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 106 | 111 | 111
Scores on a scale | -3.21 (0.27) | -5.68 (0.27) | -5.48 (0.27)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.48, 95% CI 2-sided [-3.23 to -1.73] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.27, 95% CI 2-sided [-3.03 to -1.52] — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Mean Change From Baseline in the Daily rTOSS Over the 4 Weeks Treatment Period
Description: as for outcome 4
Time Frame: Baseline and up to Week 4
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Scores on a scale | -1.41 (0.10) | -1.52 (0.10) | -1.70 (0.10)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p = 0.442, ANCOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.38 to 0.17] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p = 0.035, ANCOVA; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-0.57 to -0.02] — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Mean Change From Baseline in Rescue Loratadine Use (Mean Rescue-free Days) Over the First 4 Weeks Treatment Period
Description: as for outcome 5
Time Frame: Baseline and up to Week 4
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Days | 23.74 (0.46) | 25.62 (0.46) | 26.41 (0.46)
Statistical Analysis 1: Comparison: Placebo vs FF 55 µg QD; Test type: Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [0.60 to 3.16] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FF 110 µg QD; Test type: Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 2.67, 95% CI 2-sided [1.38 to 3.95] — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Non-SAEs During the Treatment Period
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/birth defect, other situations and is associated with liver injury or impaired liver function.
Time Frame: Up to Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Participants
  non-SAEs | 51 | 52 | 65
  SAEs | 0 | 0 | 1

12. Secondary Outcome: Number of Participants With Clinical Chemistry Values Outside the Normal Range
Description: Blood samples were collected from participants at indicated time points to evaluate clinical chemistry values outside normal range. The clinical chemistry parameters including alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST), calcium, creatinine, direct bilirubin, glucose, potassium, sodium, total bilirubin, total protein and blood urea nitrogen (BUN) with values outside normal range is presented. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Participants
  ALT; >normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  ALT; >normal range; n= 118, 118, 119 | 4 | 2 | 1
  ALT; <normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  ALT; <normal range; n= 118, 118, 119 | 2 | 3 | 2
  Albumin; >normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Albumin; >normal range; n= 118, 118, 119 | 0 | 0 | 0
  Albumin; <normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Albumin; <normal range; n= 118, 118, 119 | 4 | 1 | 1
  ALP; >normal range; n= 117, 117, 117: number analyzed (Participants) | 117 | 117 | 117
  ALP; >normal range; n= 117, 117, 117 | 18 | 21 | 22
  ALP; <normal range; n= 117, 117, 117: number analyzed (Participants) | 117 | 117 | 117
  ALP; <normal range; n= 117, 117, 117 | 1 | 0 | 0
  AST; >normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  AST; >normal range; n= 118, 118, 119 | 5 | 2 | 2
  AST; <normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  AST; <normal range; n= 118, 118, 119 | 0 | 0 | 0
  Calcium; >normal range; n= 118, 117, 116: number analyzed (Participants) | 118 | 117 | 116
  Calcium; >normal range; n= 118, 117, 116 | 0 | 0 | 4
  Calcium; <normal range; n= 118, 117, 116: number analyzed (Participants) | 118 | 117 | 116
  Calcium; <normal range; n= 118, 117, 116 | 5 | 0 | 2
  Creatinine; >normal range; n= 118, 118, 118: number analyzed (Participants) | 118 | 118 | 118
  Creatinine; >normal range; n= 118, 118, 118 | 0 | 0 | 0
  Creatinine; <normal range; n= 118, 118, 118: number analyzed (Participants) | 118 | 118 | 118
  Creatinine; <normal range; n= 118, 118, 118 | 41 | 40 | 49
  Direct bilirubin; >normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Direct bilirubin; >normal range; n= 118, 118, 119 | 2 | 0 | 2
  Direct bilirubin; <normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Direct bilirubin; <normal range; n= 118, 118, 119 | 3 | 6 | 8
  Glucose; >normal range; n= 116, 117, 117: number analyzed (Participants) | 116 | 117 | 117
  Glucose; >normal range; n= 116, 117, 117 | 8 | 5 | 5
  Glucose; <normal range; n= 116, 117, 117: number analyzed (Participants) | 116 | 117 | 117
  Glucose; <normal range; n= 116, 117, 117 | 2 | 0 | 2
  Potassium; >normal range; n= 118, 118, 115: number analyzed (Participants) | 118 | 118 | 115
  Potassium; >normal range; n= 118, 118, 115 | 0 | 1 | 2
  Potassium; <normal range; n= 118, 118, 115: number analyzed (Participants) | 118 | 118 | 115
  Potassium; <normal range; n= 118, 118, 115 | 0 | 0 | 0
  Sodium; >normal range; n= 118, 118, 116: number analyzed (Participants) | 118 | 118 | 116
  Sodium; >normal range; n= 118, 118, 116 | 0 | 0 | 0
  Sodium; <normal range; n= 118, 118, 116: number analyzed (Participants) | 118 | 118 | 116
  Sodium; <normal range; n= 118, 118, 116 | 3 | 5 | 3
  Total bilirubin; >normal range; n= 117, 118, 118: number analyzed (Participants) | 117 | 118 | 118
  Total bilirubin; >normal range; n= 117, 118, 118 | 0 | 0 | 2
  Total bilirubin; <normal range; n= 117, 118, 118: number analyzed (Participants) | 117 | 118 | 118
  Total bilirubin; <normal range; n= 117, 118, 118 | 11 | 10 | 15
  Total protein; >normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Total protein; >normal range; n= 118, 118, 119 | 0 | 1 | 4
  Total protein; <normal range; n= 118, 118, 119: number analyzed (Participants) | 118 | 118 | 119
  Total protein; <normal range; n= 118, 118, 119 | 8 | 5 | 5
  BUN; >normal range; n= 118, 118, 118: number analyzed (Participants) | 118 | 118 | 118
  BUN; >normal range; n= 118, 118, 118 | 2 | 6 | 2
  BUN: <normal range; n= 118, 118, 118: number analyzed (Participants) | 118 | 118 | 118
  BUN: <normal range; n= 118, 118, 118 | 6 | 4 | 4

13. Secondary Outcome: Number of Participants With Hematology Values Outside Normal Range
Description: Blood samples were collected from participants at indicated time points to evaluate hematology values outside normal range. The hematology parameters including basophils, eosinophils, hematocrit, hemoglobin, lymphocytes, mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes, platelet, red blood cells (RBC), total neutrophils, white blood cells (WBC) with values outside normal range is presented. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Participants
  Basophils; >normal range; n= 87, 82, 94: number analyzed (Participants) | 87 | 82 | 94
  Basophils; >normal range; n= 87, 82, 94 | 6 | 3 | 7
  Basophils; <normal range; n= 87, 82, 94: number analyzed (Participants) | 87 | 82 | 94
  Basophils; <normal range; n= 87, 82, 94 | 0 | 0 | 0
  Eosinophils; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Eosinophils; >normal range; n= 118, 119, 119 | 67 | 65 | 54
  Eosionophils; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Eosionophils; <normal range; n= 118, 119, 119 | 0 | 0 | 1
  Hematocrit; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Hematocrit; >normal range; n= 118, 119, 119 | 1 | 0 | 0
  Hematocrit; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Hematocrit; <normal range; n= 118, 119, 119 | 32 | 28 | 29
  Hemoglobin; >normal range; n= 118, 119, 118: number analyzed (Participants) | 118 | 119 | 118
  Hemoglobin; >normal range; n= 118, 119, 118 | 0 | 3 | 3
  Hemoglobin; <normal range; n= 118, 119, 118: number analyzed (Participants) | 118 | 119 | 118
  Hemoglobin; <normal range; n= 118, 119, 118 | 4 | 8 | 6
  Lymphocytes; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Lymphocytes; >normal range; n= 118, 119, 119 | 37 | 32 | 32
  Lymphocytes; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Lymphocytes; <normal range; n= 118, 119, 119 | 2 | 11 | 1
  MCH; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  MCH; >normal range; n= 118, 119, 119 | 0 | 0 | 1
  MCH; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  MCH; <normal range; n= 118, 119, 119 | 26 | 27 | 19
  MCV; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  MCV; >normal range; n= 118, 119, 119 | 0 | 0 | 0
  MCV: <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  MCV: <normal range; n= 118, 119, 119 | 33 | 34 | 27
  Monocytes; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Monocytes; >normal range; n= 118, 119, 119 | 3 | 8 | 9
  Monocytes; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Monocytes; <normal range; n= 118, 119, 119 | 1 | 2 | 3
  Platelet; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Platelet; >normal range; n= 118, 119, 119 | 45 | 33 | 40
  Platelet; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Platelet; <normal range; n= 118, 119, 119 | 0 | 0 | 0
  RBC; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  RBC; >normal range; n= 118, 119, 119 | 12 | 14 | 14
  RBC: <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  RBC: <normal range; n= 118, 119, 119 | 0 | 2 | 0
  Total neutrophils; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Total neutrophils; >normal range; n= 118, 119, 119 | 2 | 5 | 5
  Total neutrophils; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  Total neutrophils; <normal range; n= 118, 119, 119 | 30 | 27 | 23
  WBC; >normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  WBC; >normal range; n= 118, 119, 119 | 16 | 17 | 17
  WBC; <normal range; n= 118, 119, 119: number analyzed (Participants) | 118 | 119 | 119
  WBC; <normal range; n= 118, 119, 119 | 2 | 1 | 2

14. Secondary Outcome: Number of Participants With Urinalysis Values Outside Normal Range
Description: Urine parameters including urine specific gravity and urine potential of hydrogen (pH) with values outside normal range is presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Time Frame: Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Participants
  Specific gravity; >normal range; n=102, 103, 98: number analyzed (Participants) | 102 | 103 | 98
  Specific gravity; >normal range; n=102, 103, 98 | 6 | 7 | 2
  Specific gravity; <normal range; n=102, 103, 98: number analyzed (Participants) | 102 | 103 | 98
  Specific gravity; <normal range; n=102, 103, 98 | 3 | 2 | 3
  pH; >normal range; n=108, 104, 103: number analyzed (Participants) | 108 | 104 | 103
  pH; >normal range; n=108, 104, 103 | 3 | 4 | 6
  pH; <normal range; n=108, 104, 103: number analyzed (Participants) | 108 | 104 | 103
  pH; <normal range; n=108, 104, 103 | 1 | 3 | 1

15. Secondary Outcome: Number of Participants With Change From Baseline in Nasal Examination
Description: A detailed nasal examination of the mucosa, septum, secretions, nasal patency, size of any polyps and ulcers was performed at specific time points. Number of participants with improved or worsened conditions are presented. Improved condition was defined as increase in number of patencies and Worsened condition was defined as decrease in number of patencies, from Baseline to Week 4. The Baseline value for a nasal examination was the most recent recorded value for Week 4 before dosing on Day 1. Change from Baseline was defined as post-dose visit value minus Baseline value.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 120 | 119 | 119
Participants
  Nostril patent; improved | 39 | 65 | 47
  Nostril patent; worsened | 8 | 0 | 2
  Septum; improved | 1 | 2 | 2
  Septum; worsened | 0 | 0 | 2
  Mucosa oedema; improved | 21 | 43 | 48
  Mucosa oedema; worsened | 1 | 0 | 0
  Mucosa crusting; improved | 2 | 4 | 0
  Mucosa crusting; worsened | 4 | 0 | 2
  Mucosa bleeding; improved | 0 | 1 | 1
  Mucosa bleeding; worsened | 1 | 0 | 1
  Secretions; improved | 26 | 55 | 58
  Secretions; worsened | 5 | 0 | 2
  Ulcers turbinates; improved | 3 | 2 | 1
  Ulcers turbinates; worsened | 1 | 2 | 1
  Polyposis turbinates; improved | 0 | 0 | 0
  Polyposis turbinates; worsened | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital signs including SBP and DBP were measured in a semi-supine position after 5 minutes rest. The most recent recorded value for Week 4 before dosing on Day 1 was considered as Baseline value. Change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available for the specified time point were analyzed.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 118 | 117 | 117
Millimeter of mercury (mmHg)
  SBP | -1.4 (11.14) | -1.4 (8.96) | -0.1 (10.39)
  DBP | -1.1 (9.95) | 0.2 (8.91) | 0.2 (8.30)

17. Secondary Outcome: Change From Baseline in Heart Rate
Description: Vital signs including heart rate were measured in a semi-supine position after 5 minutes rest. The most recent recorded value for Week 4 before dosing on Day 1 was considered as Baseline value. Change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available for the specified time point were analyzed.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 118 | 118 | 119
Beats per minute | -0.6 (8.61) | -1.1 (12.91) | -0.4 (11.18)

18. Secondary Outcome: Change From Baseline in Temperature
Description: Vital signs including temperature were measured in a semi-supine position after 5 minutes rest. The most recent recorded value for Week 4 before dosing on Day 1 was considered as Baseline value. Change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available for the specified time point were analyzed.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 118 | 118 | 119
Degree Celsius | -0.06 (0.339) | -0.01 (0.328) | -0.01 (0.311)

19. Secondary Outcome: Change From Baseline in Respiration Rate
Description: Vital signs including respiration rate were measured in a semi-supine position after 5 minutes rest. The most recent recorded value for Week 4 before dosing on Day 1 was considered as Baseline value. Change from Baseline was defined as post-dose visit value minus Baseline value. Only those participants with data available for the specified time point were analyzed.
Time Frame: Baseline and Week 4
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
Number analyzed (Participants) | 118 | 118 | 119
Breaths per minute | 0.0 (2.51) | -0.4 (1.93) | -0.3 (1.61)

ADVERSE EVENTS:
Time Frame: On-therapy SAEs and non-SAEs are presented from the start of study treatment up to Week 4
Description: On-therapy SAEs and non-SAEs are reported for the ITT Population.
Arm/Group | Placebo | FF 55 µg QD | FF 110 µg QD
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/119 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/119 | 1/119
Other Adverse Events (participants affected / at risk) | 51/120 | 52/119 | 65/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | FF 55 µg QD (N=119) | FF 110 µg QD (N=119)
Tonsillitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=120) | FF 55 µg QD (N=119) | FF 110 µg QD (N=119)
Upper respiratory tract infection (Infections and infestations) | 15 | 26 | 19
Sinusitis (Infections and infestations) | 1 | 4 | 1
Tonsillitis (Infections and infestations) | 1 | 2 | 2
Bronchitis (Infections and infestations) | 2 | 2 | 1
Nasopharyngitis (Infections and infestations) | 0 | 3 | 2
Otitis media acute (Infections and infestations) | 3 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Myringitis (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 0
Rubella (Infections and infestations) | 0 | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Nasal mucosal erosion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
White blood cell count increased (Investigations) | 2 | 1 | 2
Blood uric acid increased (Investigations) | 1 | 1 | 0
Neutrophil percentage increased (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 0 | 1
Urobilinogen urine increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Pyrexia (General disorders) | 4 | 0 | 3
Chest discomfort (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Eschar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT02424539/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT02424539/SAP_001.pdf